CLINICAL TRIAL: NCT06586853
Title: Assessment of Complications and Outcome of Regular Hemodialysis Patients in Upper Egypt: Two Center Prospective Study
Brief Title: Outcome and Complications of Regular Hemodialysis
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohsen Abouelhassan Ramadan Sedik, Resident Doctor, Assiut University
Other Study IDs: Outcome of Hemodialysis
Record Dates: First submitted 2024-08-24; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Hemodialysis Complication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hemodialysis patients in Horus hospital: 250 patients will be studied for complications and outcome of regular hemodialysis sessions in Horus hospital
- Hemodialysis patients in Isis hospital: 50 patients will be studied for complications and outcome of regular hemodialysis sessions in Isis hospital

SUMMARY:
Assessment of the major hemodialysis outcomes which are vascular access events, mortality and hospitalization Quality of life in end stage renal disease (ESRD) patients undergoing regular hemodialysis in upper Egypt and analysis of the major hemodialysis outcomes along a one year duration.

DETAILED DESCRIPTION:
Regular dialysis treatment has been available at a national level in Egypt for more than three decades. Hemodialysis is a vital and lifesaving procedure so that many organizations, including governmental and non-governmental bodies, adopt it. Hemodialysis service is usually provided by either non-profit- or profit-based bodies.

Dialysis therapy ameliorates many of the clinical manifestations of renal failure and postpones otherwise imminent death . Despite this undeniable success, hemodialysis patients have higher mortality and hospitalization rates and lower quality of life than the general population. Also, patients must contend with unique treatment complications, such as vascular access failure, at considerable expense and morbidity .

Effective hemodialysis requires repeated and reliable access to the bloodstream through a central venous catheter or a surgically created arteriovenous communication (an autologous fistula or a synthetic graft). However, vascular access thrombosis and infection occur frequently and are the leading cause of dialysis-related morbidity.

Mortality in hemodialysis patients: The greatest number of deaths were due to infections, followed by withdrawal from dialysis, cardiac, sudden death, vascular, and other.

Quality of life in hemodialysis patients is reduced in all the health domains of Hemodialysis patients. Older age, male gender, unemployment, and duration of dialysis adversely affected the QOL scores.

Hospitalization in hemodialysis: Patients with end-stage kidney disease (ESKD) have a greater risk of comorbidities, including diabetes and anemia, and have higher hospital admission rates than patients with other diseases. The cause of hospital admissions is associated with end-stage kidney disease (ESKD) prognosis.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 18 years old.
2. Patients receiving regular maintenance hemodialysis for at least three months
3. Patients receiving regular hemodialysis (three times a week for four hours each session).
4. Patients treated at an in-center hemodialysis

Exclusion Criteria:

1. Patients treated with a home-based hemodialysis .
2. Non end stage renal disease patients undergoing hemodialysis due to any other indication.
3. Refuse to share in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic kidney disease on regular hemodialysis with age more than 18 years old in 2 dialysis centers in Upper Egypt
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of the major hemodialysis outcomes | 3 months
  Assessment of the major hemodialysis outcomes including change in serum creatinine in mg\dl

CONTACTS AND LOCATIONS:
Overall Officials: Mohsen A Ramadan, Master, Principal Investigator — Assiut University; Samir k Abdelhamid, professor, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zhao X, Niu Q, Gan L, Hou FF, Liang X, Ni Z, Chen Y, Zhao J, Bieber B, Robinson B, Chen X, Zuo L. Baseline data report of the China Dialysis Outcomes and Practice Patterns Study (DOPPS). Sci Rep. 2021 Jan 13;11(1):873. doi: 10.1038/s41598-020-79531-4. PMID 33441625
- [Background] Matsuzawa R, Kamitani T, Roshanravan B, Fukuma S, Joki N, Fukagawa M. Decline in the Functional Status and Mortality in Patients on Hemodialysis: Results from the Japan Dialysis Outcome and Practice Patterns Study. J Ren Nutr. 2019 Nov;29(6):504-510. doi: 10.1053/j.jrn.2018.10.012. Epub 2018 Dec 24. PMID 30591357